CLINICAL TRIAL: NCT04303520
Title: A Phase I Clinical Trial of T-Cells Targeting CD19 and CD22 for Subjects With CD19-positive Acute Lymphoblastic Leukemia
Brief Title: Anti-CD19/CD22 Bispecific CAR-T Cell Therapy for CD19-positive ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Collaborators: Hrain Biotechnology Co., Ltd. (Industry); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-CD19/CD22 CAR-T
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: CD19-positive ALL
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/CD22 CAR-T cells (Experimental): Administration with anti-CD19/CD22 CAR-T cells in the CD19-positive ALL patients
  Interventions: Biological: anti-CD19/CD22 CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19/CD22 CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-CD19 and anti-CD22 CARs
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 500mg/m2/d

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-CD19/CD22 bispecific chimeric antigen receptors (CARs) T cell therapy for CD19-positive Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the feasibility ad safety of anti-CD19/ CD22 CAR-T cells in treating patients with CD19-positive Acute Lymphoblastic Leukemia.

Secondary Objectives

1. To determine in vivo expression, dynamics and persistency of anti-CD19/CD22 CAR-T cells.
2. To determine in vivo expression of CD19-positive B cells.
3. To access the complete remission rate (ORR) in patients with ALL with 3 months after CD19/CD22 CAR-T cells infusion.
4. To investigate the favorable CD19/CD22 CAR-T cells dose and dosage regimen for the Phase II Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

1. 13 Years to 70 Years, Male and female;
2. Expected survival > 12 weeks;
3. Clinical performance status of ECOG score 0-2;
4. Histologically confirmed as CD19-positive lymphoma and who meet one of the following conditions:

   * Patients received at least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment;
   * Disease recurrence after stem cell transplantation.
5. Accessible to intravenous injection, and no white blood cell collection contraindications
6. Patients who meet the following conditions:

   * Creatinine < 2.5 mmol/l;
   * Cardiac ejection fraction>50%, no pericardial effusion and no pleural effusion (ECHO examination);
   * Baseline oxygen saturation>92%;
   * Total bilirubin≤1.5xULN;
   * ALT/AST≤2.5x normal.
7. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. Accompanied by other malignant tumor
2. Active hepatitis B, hepatitis C, syphilis, HIV infection
3. Suffering severe cardiovascular or respiratory disease
4. Any other diseases could affect the outcome of this trial
5. Any affairs could affect the safety of the subjects or outcome of this trial
6. Pregnant or lactating women, or patients who plan to be pregnancy during or after treatment
7. Occurrence of infection uncontrolled or requiring systemic treatment 14 days prior to assignment
8. Patients who are accounted by researchers to be not appropriate for this test
9. Received CAR-T treatment or other gene therapies before assignment
10. Patients with symptoms of central nervous system
11. Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 6 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 8 weeks
  Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm
Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation
Total number of CAR-positive T cells infiltrated into lymphoma tissue | 6 months
  Total number of CAR-positive T cells infiltrated into lymphoma tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Province of TCM, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Litzow MR. Hematology clinic. Acute lymphoblastic leukemia. Hematology. 2014 Jun;19(4):246-7. doi: 10.1179/1024533214Z.000000000281. No abstract available. PMID 24856441
- [Background] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Background] Bhojwani D, Pui CH. Relapsed childhood acute lymphoblastic leukaemia. Lancet Oncol. 2013 May;14(6):e205-17. doi: 10.1016/S1470-2045(12)70580-6. PMID 23639321
- [Background] Raetz EA, Bhatla T. Where do we stand in the treatment of relapsed acute lymphoblastic leukemia? Hematology Am Soc Hematol Educ Program. 2012;2012:129-36. doi: 10.1182/asheducation-2012.1.129. PMID 23233571
- [Background] Uckun FM, Jaszcz W, Ambrus JL, Fauci AS, Gajl-Peczalska K, Song CW, Wick MR, Myers DE, Waddick K, Ledbetter JA. Detailed studies on expression and function of CD19 surface determinant by using B43 monoclonal antibody and the clinical potential of anti-CD19 immunotoxins. Blood. 1988 Jan;71(1):13-29. PMID 3257143
- [Background] Onea AS, Jazirehi AR. CD19 chimeric antigen receptor (CD19 CAR)-redirected adoptive T-cell immunotherapy for the treatment of relapsed or refractory B-cell Non-Hodgkin's Lymphomas. Am J Cancer Res. 2016 Jan 15;6(2):403-24. eCollection 2016. PMID 27186412
- [Background] Ramos CA, Heslop HE, Brenner MK. CAR-T Cell Therapy for Lymphoma. Annu Rev Med. 2016;67:165-83. doi: 10.1146/annurev-med-051914-021702. Epub 2015 Aug 26. PMID 26332003
- [Background] Gardner RA, Finney O, Annesley C, Brakke H, Summers C, Leger K, Bleakley M, Brown C, Mgebroff S, Kelly-Spratt KS, Hoglund V, Lindgren C, Oron AP, Li D, Riddell SR, Park JR, Jensen MC. Intent-to-treat leukemia remission by CD19 CAR T cells of defined formulation and dose in children and young adults. Blood. 2017 Jun 22;129(25):3322-3331. doi: 10.1182/blood-2017-02-769208. Epub 2017 Apr 13. PMID 28408462
- [Background] Turtle CJ, Hanafi LA, Berger C, Gooley TA, Cherian S, Hudecek M, Sommermeyer D, Melville K, Pender B, Budiarto TM, Robinson E, Steevens NN, Chaney C, Soma L, Chen X, Yeung C, Wood B, Li D, Cao J, Heimfeld S, Jensen MC, Riddell SR, Maloney DG. CD19 CAR-T cells of defined CD4+:CD8+ composition in adult B cell ALL patients. J Clin Invest. 2016 Jun 1;126(6):2123-38. doi: 10.1172/JCI85309. Epub 2016 Apr 25. PMID 27111235
- [Background] Park JH, Geyer MB, Brentjens RJ. CD19-targeted CAR T-cell therapeutics for hematologic malignancies: interpreting clinical outcomes to date. Blood. 2016 Jun 30;127(26):3312-20. doi: 10.1182/blood-2016-02-629063. Epub 2016 May 20. PMID 27207800
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Derived] Ma Q, Wei R, Wang Q, Jiang S, Wu Y, Min C, Guo S, Zhang Y, Sun X, Wu H, Sun X, Xiang F, Xiao M, Cheng Z. A bi-specific CAR-T cell therapy targeting CD19 and CD22 in relapsed or refractory B-ALL. Clin Exp Med. 2025 Jul 28;25(1):264. doi: 10.1007/s10238-025-01637-8. PMID 40719826